CLINICAL TRIAL: NCT05812599
Title: Rapid Acceleration of Diagnostics Underserved Populations Supplement: Understanding COVID-19 Testing Knowledge and Practices Among 2-1-1 Helpline Callers
Brief Title: Understanding COVID-19 Testing Knowledge and Practices Among 2-1-1 Helpline Callers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Matthew Kreuter, Principal Investigator, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 3R01CA235773-03S1 (NIH)
Record Dates: First submitted 2022-11-29; First posted 2023-04-13 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Communication; Health Knowledge, Attitudes, Practice
MeSH Terms: conditions — Communication; Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COVID Test Learning Module (Experimental): In the experimental condition, participants will respond to survey questions (pre-exposure) before being presented with four narrative scenarios, questions, and accompanying messages about COVID testing (exposure), followed by post-test survey questions about COVID testing behaviors (post-exposure).
  Interventions: Other: Educational Module
- Control (No Intervention): In the control condition, participants will respond to survey questions (pre-exposure) and post-test survey questions about COVID testing behaviors (post-exposure) only.

INTERVENTIONS:
Other: Educational Module — The COVID Test Learning Module will present four multi-part character scenarios that someone might experience when considering testing for COVID-19. Participants will answer questions about the character's behavior. Accurate guidelines will be provided in response to each scenario to educate participants about what to do in nuanced COVID testing decision-making situations.
  Arms: COVID Test Learning Module

SUMMARY:
The purpose of this study is to identify promising health education strategies and culturally appropriate messages for use by 2-1-1 practitioners to promote coronavirus disease of 2019 (COVID) testing behaviors. Previous study findings and evidence-based health communication and education tactics were integrated to create an interactive learning module that includes four narrative scenarios, illustrations, and accompanying questions and responses that inform the audience about COVID testing guidelines. The study will test the effectiveness of the interactive learning module with 2-1-1 callers (n=300) in Connecticut, North Carolina, and Nebraska. Participants' contact information will be shared with us by 2-1-1 with the participants' given consent. The study team will send the potential participant via text message a link to a survey that includes a screen where they will provide informed consent. Those who provide consent will be randomly assigned to receive one of two surveys. The inclusion of the interactive learning module is what varies across the surveys. An experimental group will receive the learning module with a study team-developed pre- and post-survey, and the control group will receive only the study team-developed pre- and post-survey. The post-survey contains questions regarding information covered in the interactive learning module. It is hypothesized that those who complete the interactive learning module in the experimental group will score better on the post-survey questions when compared to the control group. All participants, regardless of experimental or control condition, will receive an information sheet with the most up-to-date scientific guidelines for COVID testing.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who called 211 in Connecticut, Nebraska, or North Carolina on behalf of themselves or their families
* Must be 18 or older
* Must have English language proficiency
* Must be willing to be contacted via text messages or email

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 298 (Actual)
Dates: Start 2022-09-22 (Actual); Primary Completion 2023-01-20 (Actual); Study Completion 2023-01-20 (Actual)

PRIMARY OUTCOMES:
Proportion of participants who answer post-test questions correctly | Through survey completion, an average of 10-15 minutes.
  The primary objective of this study is to evaluate differences in knowledge regarding COVID testing between 2-1-1 callers randomized to the control vs. experimental group. Participants who do better would answer more items correctly on the COVID prevention knowledge post-test. Assessed using a non-parametric t-test.

SECONDARY OUTCOMES:
Number of participants with knowledge gained after exposure to learning module | Through survey completion, an average of 10-15 minutes.
  A secondary outcome is to identify if exposure to the learning module increased participant knowledge about COVID prevention. Assessed by comparing the percentage of correct answers from questions within the learning module to the percentage of correct answers in the post-test.

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University in St. Louis, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided